CLINICAL TRIAL: NCT02108665
Title: Magnetic Resonance Imaging Hysterosalpingography Versus Radiographic Hysterosalpingography in Female Infertility
Brief Title: Magnetic Resonance Imaging (MRI) Hysterosalpingography Versus Radiographic Hysterosalpingography in Female Infertility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 11AOI07
Record Dates: First submitted 2014-04-07; First posted 2014-04-09 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2017-10

CONDITIONS: Female Infertility
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Radiographic hysterosalpingography (Other): Realisation in first: radiographic hysterosalpingographyresonance then imaging hysterosalpingography
  Interventions: Radiation: Radiographic hysterosalpingography; Radiation: Magnetic resonance imaging hysterosalpingography
- Magnetic resonance imaging hysterosalpingography (Other): Realisation in first : magnetic resonance imaging hysterosalpingography then a radiographic hysterosalpingography
  Interventions: Radiation: Radiographic hysterosalpingography; Radiation: Magnetic resonance imaging hysterosalpingography

INTERVENTIONS:
Radiation: Radiographic hysterosalpingography
Radiation: Magnetic resonance imaging hysterosalpingography

SUMMARY:
The main objective of this study is to compare the data of Hystérosalpingo-MRI with intra cavitary injection of diluted gadolinium salts with the classic hysterography, which allows to realize at once with no irradiating examination, a complete assessment of the female infertility.

DETAILED DESCRIPTION:
Infertility is a disease which affects around 15% of couples (one union of seven) and has been increasing for 10 years. Therefore, and due to the development of methods of medically assisted procreation, demand for infertility evaluation is steadily increasing.

The infertility evaluation always begins with an accurate history, coupled with a physical examination of both partners. Indeed, infertility of a couple is due to the female partner in about two thirds of cases, the male partner in the remaining third of cases. In women, the main observed causes are ovulatory function disorders (10 to 20%), tubal causes by proximal or distal occlusion (10%), uterine causes involving intra-uterine synechiae, leiomyomas, adenomyosis, mucosal polyps (5 %), inadequate cervical mucus or cervical stenosis , and peritoneal causes such as endometriosis and post-infectious or post-surgical peritubo-ovarian adhesions (20 %).

Medical imaging is one of the key methods to identify the different etiologies in men as in women. It will serve to clarify the etiology in question and assess the likelihood of subsequent pregnancy. The initial imaging assessment for infertility in any woman includes an endovaginal ultrasound examination and a hysterosalpingography (HSG) . The use of MRI is considered as a second line in the absence of definitive diagnosis or to establish a definitive diagnosis before considering a targeted therapy. Indeed the performance of MRI for the diagnosis of pelvic endometriosis or fibroids mapping are well established.

HSG is the imaging technique of choice to evaluate the morphology of the uterine cavity and tubal patency. But it has several important limitations. Firstly it is an imaging method that uses x-rays and therefore delivers irradiation to the gynecological organs. Moreover, it does not allow a precise exploration of the entire abdomen and pelvis: therefore, the physician cannot have a complete assessment of the etiologies of infertility with HSG. Finally, it has a very good specificity but a relatively low sensitivity.

ELIGIBILITY:
Inclusion Criteria:

Patient who a pelvic MRI and an Hysterography, part of an infertility assessment, have been prescribed by a gynecologist physician in Nice University Hospital.

Informed consent signed Patient with social insurance Age > 18

Exclusion Criteria:

Contraindication to magnetic resonance imaging hysterosalpingography Contraindication to radiographic hysterosalpingography

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Diagnostic performance of hystérosalpingo-MRI | one day
  To assess the diagnostic performance of hystérosalpingo-MRI by its sensitivity, specificity, negative predictive value, positive predictive value.
  To determine uterine cavity abnormality by the presence of the following abnormalities: synechiae, polyp, intra cavitary myoma, adenomyosis, uterine malformation.

CONTACTS AND LOCATIONS:
Overall Officials: Madleen CHASSANG, MD, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- Service d'imagerie médicale Hôpital Archet II, Nice, France